CLINICAL TRIAL: NCT06886204
Title: Youth Participatory Action Research to Prevent Community Violence Among Black Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Briana Woods-Jaeger, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006694; R01CE003580 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Community Violence
Keywords: Youth Participatory Action Research; Youth Empowered Advocating for Health; Community violence
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YEAH group: Immediate Intervention (Other): YEAH is a YPAR intervention that involves conducting a photovoice project to explore youth perspectives on the structural determinants of community violence and developing a theater performance to share the key themes and action priorities generated from photovoice with youth and adults in their community.
  The team will conduct individual-level surveys at baseline, 8 weeks, and 3 months to assess individual-level impacts of YEAH on youth participants
  Interventions: Behavioral: YEAH: Youth Empowered Advocating for Health
- YEAH group: Delayed (Other): Youth who are randomized to waitlist control will be offered the 8-session YEAH intervention after data collection is complete with the YEAH immediate intervention group
  Interventions: Behavioral: YEAH: Youth Empowered Advocating for Health

INTERVENTIONS:
Behavioral: YEAH: Youth Empowered Advocating for Health — The Youth Empowered Advocating for Health (YEAH) program is a Youth Participatory Action Research (YPAR) intervention aimed at addressing community violence by fostering youth and community healing. It combines photovoice and theater arts performances.
  In photovoice sessions, Black youth explore structural determinants of community violence through a participatory research process. Guided by trained facilitators, youth learn the method after obtaining parental consent and youth assent. Using the structured SHOWED framework, they analyze and discuss images, generating ideas for social action. During the photovoice sessions, photo assignments will be completed, with discussions recorded, analyzed for themes, and shared for validation.
  The final four sessions will integrate these themes into theater arts performances, allowing youth to creatively express insights and experiences, fostering empowerment and social change.
  Other Names: YEAH

SUMMARY:
This behavioral intervention study aims to evaluate the effectiveness of Youth Empowered Advocating for Health (YEAH) on youth prosocial behavior and aggressive behavior and assess racial identity and future orientation as mediators of prevention effects.

DETAILED DESCRIPTION:
Structural determinants of violence such as residential segregation, concentrated poverty, and limited access to education and employment, disproportionately affect Black youth. This group subsequently faces the highest rates of violence exposure and related injuries, with homicide being a leading cause of death. In addition, the consequences of violence exposure include academic decline, psychological issues, and chronic health conditions.

It is important to address the long-lasting effects of structural violence among Black youth including emotional distress and eroding family and community ties. Current violence prevention methods often overlook the impact of structural violence.

The proposed solution is a Youth Participatory Action Research (YPAR) intervention, called Youth Empowered Advocating for Health (YEAH), which aims to empower Black youth and improve their outcomes. The YEAH program, developed over ten years in partnership with youth, focuses on empowering youth to explore topics of concern in their community and generate solutions. This study will evaluate YEAH's effectiveness in reducing community violence in Metro Atlanta, emphasizing community healing and empowerment as well as narrative change as vital strategies for prevention.

ELIGIBILITY:
Inclusion Criteria:

* Identify their race or ethnicity as Black or African American
* Speak English
* Able to understand the project and give full consent to participate if eligible
* Have a parent or guardian provide consent for them to participate
* Member of Boys and Girls Clubs or other Youth Serving Organization (YEAH immediate intervention and delayed intervention groups)

Exclusion Criteria:

* Non-English speakers

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in prosocial behavior: Multidimensional Well-being Assessment Scale | Baseline, Week 8, Month 3
  Youth prosocial behavior will be measured using a scale developed by Grills et al. (2016) which assesses youth endorsement of behaviors that build connections with others in the past 2 weeks (α=.92). This 12-item scale was developed from items from the Multidimensional Well-being Assessment Scale, and uses a Likert-type scale (1=never; 5=always), with higher mean scores indicating greater likelihood of engaging in behaviors that reflect care and concern for others
Change in aggressive behavior: California Healthy Kids Survey adaptation | Baseline, Week 8, Month 3
  Youth aggressive behavior will be measured using 10 items adapted from the California Healthy Kids Survey. This measure asks participants how often they engaged in behaviors such as yelling at teachers, hitting or punching someone, or teasing another student in the past month (α=.88). These items assess the frequency of behaviors with 5 response categories (0,1,2,3,4+).
Change in community violence exposure: Community Experiences Questionnaire | Baseline, Week 8, Month 3
  This will be measured with 14 items (items 12-25) from the Community Experiences Questionnaire assessing exposure to violence by witnessing (CEQ-WIT). This scale asks the respondent to rank the frequency with which they have experienced each item on a 4-point rating scale (1=never, 2=once, 3=a few times, 4=lots of times). Scores are calculated by averaging respondents' ratings for the scale

SECONDARY OUTCOMES:
Racial identity: multidimensional inventory of Black identity-teen (MIBI-T)score | Baseline, Week 8, Month 3
  Racial identity will be measured using the multidimensional inventory of Black identity-teen (MIBI-T), including centrality, private regard, public regard, nationalism, humanism, assimilation, and oppressed minority. The scale includes 21 items on a Likert-type scale (1=really disagree; 5=agree), with higher mean scores indicating more positive racial identity
Future orientation: Hemingway Measure of Adolescent Connectedness | Baseline, Month 3
  This will be measured using 4 items selected from the Hemingway Measure of Adolescent Connectedness as used by Grills et al. (2016). These items assess participants' orientation toward the future by rating their expectations and aspirations on a 5-point Likert-type scale (1=strongly disagree; 5=strongly agree), with higher scores indicating more positive expectations for the future (α=.84).

CONTACTS AND LOCATIONS:
Overall Officials: Briana Wood-Jaeger, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Boys & Girls Club of Metro Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request with data use agreements in place
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: May 2028 onwards
Access Criteria: Emory Dataverse